CLINICAL TRIAL: NCT00479752
Title: A Randomized, Open-label Phase II Study Evaluating the Efficacy and Safety of FOLFOX4 + Weekly Cetuximab Versus FOLFOX4+ Biweekly Cetuximab as First-line Therapy in Patients With Metastatic Colorectal Cancer.
Brief Title: Safety and Efficacy of Folfox4 + Weekly Cetuximab vs Folfox 4+Biweekly Cetuximab by Metastatic Colorectal Cancer
Acronym: CORE 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Central European Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CECOG /CORE 1.2.002
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): FOLFOX4:
  * Oxaliplatin 85 mg/m² d1
  * Leucovorin 200 mg/m² d1+d2, followed by
  * Bolus 5FU 400 mg/m², followed by
  * Infusional 5FU 600 mg/m²,over 22 hours, every 2 weeks
  Cetuximab is administered to arm A of the study as an infusion with initial dose 400 mg/m² in week 1 followed by weekly doses of 250 mg/m².
  Interventions: Drug: FOLFOX4 (Oxaliplatin), Cetuximab
- B (Active Comparator): FOLFOX4:
  * Oxaliplatin 85 mg/m² d1
  * Leucovorin 200 mg/m² d1+d2, followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 600 mg/m², over 22 hours, every 2 weeks
  Cetuximab is administered to arm B of the study as infusions of 500 mg/m² every two weeks.
  Interventions: Drug: FOLFOX4 (Oxaliplatin), Cetuximab

INTERVENTIONS:
Drug: FOLFOX4 (Oxaliplatin), Cetuximab — Arm A FOLFOX4:
  * Oxaliplatin 85 mg/m² d1
  * Leucovorin 200 mg/m² d1+d2, followed by
  * Bolus 5FU 400 mg/m², followed by
  * Infusional 5FU 600 mg/m²,over 22 hours, every 2 weeks
  Cetuximab is administered to arm A of the study as an infusion with initial dose 400 mg/m² in week 1 followed by weekly doses of 250 mg/m².
  Arm B FOLFOX4:
  * Oxaliplatin 85 mg/m² d1
  * Leucovorin 200 mg/m² d1+d2, followed by
  * Bolus 5FU 400 mg/m² , followed by
  * Infusional 5FU 600 mg/m², over 22 hours, every 2 weeks
  Cetuximab is administered to arm B of the study as infusions of 500 mg/m² every two weeks.

SUMMARY:
To assess the efficacy of FOLFOX4 in combination with cetuximab, weekly and FOLFOX4 in combination with cetuximab, biweekly.

DETAILED DESCRIPTION:
This multicenter randomized phase II study will enroll approximately 150 patients with metastatic Colorectal Cancer. Patients are randomized in Arm A(FOLFOX4 in combination with weekly Cetuximab) or Arm B (FOLFOX4 in combination with biweekly Cetuximab). Both efficacy and safety data will be collected. The investigator will assess response to treatment every 8 weeks based on the imaging.

Following permanent treatment cessation, patients will be followed-up for survival.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female ≥ 18 years of age
* Diagnosis of histologically confirmed adenocarcinoma of the colon or rectum
* Metastatic colorectal carcinoma not suitable for curative-intent resection- Availability of tumor sample (or able and willing to provide tumor sample) for EGFR assessment
* Presence of at least one lesion measurable unidimensionally by CT scan or MRI. (Target lesion(s) must not lie within an irradiated area)
* Karnofsky performance status of > 80 at study entry
* Leucocytes ≥ 3.0 x 10 9/L and neutrophils ≥1.5 x 10 9/L, platelets ≥ 100 x 10 9/L, and hemoglobin ≥ 9 g/dL.
* Bilirubin ≥ 1.5 x ULN
* ASAT and ALAT ≤ 2.5 x ULN (≤5 x ULN if liver metastasis are present)
* Serum creatinine ≤ 1.5 x ULN

Exclusion Criteria:

* Brain metastasis (known or suspected)
* Previous chemotherapy for metastatic disease. Prior adjuvant chemotherapy is allowed if the chemotherapy treatment free interval is > 6 months.
* Surgery (excluding diagnostic biopsy) or irradiation within 4 weeks prior to study entry
* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Any investigational agent(s) within 4 weeks prior to entry
* Previous exposure to EGFR-pathway targeting therapy
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 12 months
* Acute or subacute intestinal occlusion or history of inflammatory bowel disease
* Pre-existing neuropathy > grade 1. In case of prior oxaliplatin containing adjuvant chemotherapy: pre-existing neuropathy ≥ 1.
* Known grade 3 or 4 allergic reaction to any of the components of the treatment.
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 5 years will be allowed to enter the trial)
* Pregnancy or lactation
* Inadequate contraception (male or female patients) if of childbearing or procreational potential
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the trial is: • Objective response (CR/PR), as assessed by RECIST criteria | The objective response rate - defined as the rate of subjects with complete response (CR) or partial response (PR)
  Objective response (partial or complete) will be assessed using RECIST criteria. The objective response rate (defined as the rate of subjects with complete response (CR) or partial response (PR)) will be estimated and associated exact two-sided 95% confidence limit (Clopper-Pearson) will be calculated. In addition to the estimates within each treatment group odds ratios and associated 95% CI will be calculated using the Cochran Mantel-Haenszel procedure.

SECONDARY OUTCOMES:
• Progression Free Survival (PFS) • Overall survival • Safety/Adverse events Safety | he rate of subjects with complete response (CR) or partial response (PR)
  Secondary objectives are the estimation of differences in PFS and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Tudor Ciuleanu, Prof. Dr., Principal Investigator — Institutul Oncologic of Cluj
Locations (24):
- Austria (2):
  - LKH Leoben, Abt. für Innere Medizin, Leoben, Styria
  - Medical University of Vienna, Vienna
- Institute of Oncology Sarajevo, Sarajevo, Bosnia and Herzegovina
- SBALO National Oncology Center, Sofia, Bulgaria
- Croatia (3):
  - University Hospital Centre Rijeka, Rijeka
  - University Hospital for Tumors, Zagreb
  - University Hospital Rebro, Zagreb
- Noth estonian Regional Oncology Hospital, Tallinn, Estonia
- Greece (2):
  - AHEPA Hospital University Hospital Papageorgiou, Athens
  - General Hospital of Athens, Athens
- Hungary (3):
  - Semmelweis Univ. Radiology Clinic, Budapest
  - National Medical Center, Budapest
  - Markusovsy Hospital, Szombathely
- Israel (2):
  - Meir Medical Center, Kfar Saba
  - Oncology Division Sourasky Medical Center, Tel Aviv
- Latvia (2):
  - P. Stradins University Hospital, Riga
  - latvian Center of Oncology, Riga
- Romania (2):
  - Institutul Oncologic Bucuresti, Bucharest
  - Institutul Oncologic Ion Chiricuta, Cluj-Napoca
- Serbia (2):
  - Institute of Oncology and Radiology of Serbia, Belgrade
  - Institute of Oncology of Vojvodina, Kamenitz
- Slovakia (2):
  - National Cancer Institute, Bratislava
  - National Institute of Oncology, Bratislava
- Institute of Oncology, Ljubljana, Slovenia